CLINICAL TRIAL: NCT03841669
Title: Behavioral Studies of Cardiovascular Disease
Brief Title: Exercise, Brain, and Cardiovascular Health
Acronym: eBACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kirk Erickson, PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY19020218; P01HL040962 (NIH)
Record Dates: First submitted 2019-01-22; First posted 2019-02-15 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases
Keywords: Brain; Cardiovascular Disease; Exercise; Brain Health
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 130 individuals between the ages of 26 and 58 will be randomly assigned to one of two groups; Aerobic Exercise group or Physical Activity and Health Information group. The exercise group will receive moderate to vigorous intensity aerobic exercise targeting 150 minutes per week for 12 months. The group will target dividing these minutes into 3 exercise sessions a week over a 12-month period. Both groups will be asked to wear activity monitors every 6 weeks. Both groups will have fitness testing and cardiovascular assessments completed at baseline, 6 months (optional) and following the completion of the 12-month intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Neither the investigator, nor outcomes assessors will know participants' group assignment. Participants will be instructed to refrain from speaking about their group's activities when visiting the lab for 6 month (if applicable) and follow-up assessments.In addition, special care was taken to ensure that non-blinded laboratory staff (i.e. staff member notifying participants of their group assignments, staff monitoring the intervention) are not located in the same proximity in the laboratory, further preventing accidental unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Group (Experimental): This is the experimental group. Exercise is prescribed for 150 min/week. Due to COVID-19 restrictions the exercise supervision was allowed to be either remotely or in the context of a laboratory setting.
  Interventions: Behavioral: Aerobic Exercise Group
- Physical Activity & Health Information Group (Active Comparator): This is the control group. Participants will engage in daily life monitoring every 6 weeks.
  Interventions: Behavioral: Physical Activity & Health Information Group

INTERVENTIONS:
Behavioral: Aerobic Exercise Group — Guidelines for exercise programming (ACSM, 2018) will be followed including a warm up and cool down, progressive and gradual increments in duration, and instruction regarding avoidance of physical activity related injury. The exercise group will receive moderate to vigorous intensity aerobic exercise targeting 150 minutes per week for 12 months. The group will target dividing these minutes into 3 exercise sessions a week. The prescribed intensity will be based on their maximal fitness testing heart rate and then calculated per a research grade method. They will maintain a minimum heart rate from their specific calculation that will be monitored by Polar Heart Rate straps.
  Arms: Aerobic Exercise Group
Behavioral: Physical Activity & Health Information Group — This group will not partake in the aerobic fitness sessions but will be asked to wear a daily monitoring device every 6 weeks. They will also complete all baseline, 6-month (optional), and 12-month visits.
  Arms: Physical Activity & Health Information Group

SUMMARY:
eBACH is a randomized intervention to determine the effects of aerobic exercise on brain structure and function, as well as to determine how exercise-induced training effects relate to cardiovascular function via related brain changes.

DETAILED DESCRIPTION:
Aim 1: To determine the neurobiology of exercise and cardiovascular factors: (1A) Body- to -Brain hypothesis: Exercise -induced changes in peripheral markers of cardiovascular health (e.g., cardiorespiratory fitness, peripheral vascular function) will precede and partly explain (statistically mediate) some of the exercise -induced changes in functional and structural features of areas defining visceral control circuits. (1B) Brain- to -Body hypothesis: Exercise -induced changes in functional and structural features of areas defining visceral control circuits precede and partly explain (statistically mediate) consequent changes in autonomic and neuroendocrine mediators of cardiovascular function that are under neural regulation, including baro-reflex sensitivity and heart rate variability. Aim 2: To determine the neurobiology of exercise self--reported correlates of cardiovascular function: (2A) Exercise will induce changes in visceral control areas engaged by functional magnetic resonance imaging (fMRI) tasks, and these changes will partly explain exercise- induced reductions in cardiovascular responsivity to challenges in daily life. (2B) Exercise will induce changes in visceral control areas engaged by an functional magnetic resonance imaging (fMRI) emotion processing and regulation paradigm, and these changes will partly explain exercise- induced improvements in affect measured in daily life by EMA and by conventional self- report instruments. The public health significance of this research is that it is designed to more precisely define and refine neurobiological targets to improve cardiovascular function and health.

Because of disruptions due to COVID-19, the study was placed into a compromised position that required conservation of funds and resources, resulting in a narrowing of focus and an abbreviated assessment protocol that limited the scale and scope of the longitudinal assessments and also reduced the sample size. As such, several of the secondary outcomes that were pre-specified were moved to "other pre-specified" during the course of the project.

ELIGIBILITY:
Inclusion Criteria:

* Age - individuals aged 26-58 years old
* Gender & Ethnicity - men and women are both eligible to participate. The eBACH study expects the study population to be approximately 50% women. All ethnic groups are eligible for the study. The eBACH study expects the study population to be approximately 30% minorities.
* Ambulation - study participants must be able to walk without pain or use of an assisted walking device. This will be determined during the initial phone screen. Ambulation will also be assessed in person as the potential subject must be able to complete the VO2 Max test on a treadmill.
* Physical Activity Level - all participants must exercise less than 100 minutes per week and have a VO2max percentile level less than 75 based on the ACSM Guidelines for Exercise Testing (9th and 10th edition).
* Residency - Since the intervention is 12 months in duration, all potential participants must reside in the Pittsburgh area and plan on residing in the area for at least one year after randomization. It is recommended that the study coordinator during the second screen assess potential participants' distance from the exercising sites since the study requires 2 visits per week. The further a participant is from an intervention site, the higher the probability they will be unable to adhere to the protocol. In addition, participants must have reliable transportation to complete the outcome measures and the intervention requirements. Questions related to these considerations are asked during the phone screen and should also be assessed during the baseline visits.
* Willingness to be randomized - To be eligible, all potential study participants must be willing to be randomized to either of the intervention arms. Individuals that insist on participating only if they can choose which arm they belong to should not be enrolled.

Exclusion Criteria:

* Current use of prescribed blood pressure medication - participants who regularly use blood pressure medication will be excluded from the study.
* Self-reported chronic psychotic illness (schizophrenia, bipolar disorder) or neurological disorder (Parkinson's disease, dementia, MCI) - the eBACH study will exclude anyone who self-reports that they experience schizophrenia, bipolar disorder or parkinson's, dementia, or mild cognitive impairment.

  * Regular use of psychotropic medications - participants who regularly use psychotropic medications is defined as taking more than 7 times in a two week period will be excluded from the study (SSRIs are permitted)
* Current pregnancy or plans to become pregnant over the next year - any woman who is pregnant via the pregnancy test at the baseline visit will be excluded from the study. A pregnancy test will also be given at the MRI visit and this will be repeated at 6-months (if applicable) and 12-months.
* Self-reported prior heart attack, stroke, bypass surgery, angioplasty, congestive heart failure, arrhythmia (cardiac rhythm problems) - any person that reports that they have any of the health conditions listed above will be excluded from the study.
* Severe hypertension (sbp/dbp greater than/or equal to 160/100)

  * >140/90 IS ALLOWED, but feedback card and information about elevated levels will be provided to the participant.
* Cancer - potential participants who have received treatment in the last 12 months for cancer, including radiation or chemotherapy will be excluded from the study. Although, if a potential participant who had non-melanoma skin cancer will be allowed to enroll in eBACH.
* Liver disease - any person who has had hepatitis B or C, liver failure or Cirrhosis will be excluded from the study.
* Kidney disease - potential participants who indicated they have chronic kidney failure, have undergone dialysis, or have had a kidney transplant will not be eligible to participant in the eBACH study.
* Type 1 diabetes and/or insulin treatment

  * Type 2 diabetics if they are taking insulin or 2 or more diabetes medications. Single injections that contain 2+ drugs count as 2 medications.
* Lung disease requiring drug treatment (any medication usage 3x/week in the last 2 weeks for chronic obstructive pulmonary disease (COPD), emphysema, asthma)

  * Rescue inhalers are okay.
* Non fluency in English - speaking/reading English everyday for <10 years
* Nightshift work - the eBACH study for the purposes of the EMA monitoring will exclude any participants who work more than 12 night shifts in the last year, or participants who work more than one night shift per month on average. This is defined as a period of work in which half or more of the hours worked are between midnight and 8:00 in the morning.
* MRI incompatable

  * Certain medical devices, implants or other metal objects in or on the body that cannot be removed and are MRI incompatible
  * Inability to fit into the MRI scanner
  * Colorblindness
  * History of injury with metal object, metal in eye, welding or working in close proximity to welding without X-ray to prove lack of metal in the body.
* Suspected alcohol use disorder - for the eBACH study alcohol use disorder is defined as having five or more drinks at one time three times or more per week.
* Those who are otherwise unable to meet the requirements of the study (persons whose employment or personal situation will not permit momentary interruptions required for electronic diary and ambulatory data)

Ages: 26 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2024-02-03 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk I Erickson, PhD, Principal Investigator — University of Pittsburgh; Peter Gianaros, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The data from this study will be made available to outside investigators under a data-sharing agreement. The data will be available to outside investigators after publication of the primary aims and at completion of quality control assessments and data organization. The investigators expect that the data from this study will result in interest from internal and external investigators for secondary analysis and ancillary projects.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Will be made available after study investigators have published summary data and primary aims results. Will be available for unlimited amount of time.
Access Criteria: Data requests will be approved by the PI and Co-PI. Requests can be made by contacting the study coordinator.

REFERENCES:
- [Derived] Molina Hidalgo C, Collins AM, Crisafio ME, Grove G, Kamarck TW, Kang C, Leckie RL, MacDonald M, Manuck SB, Marsland AL, Muldoon MF, Rasero J, Scudder MR, Velazquez-Diaz D, Verstynen T, Wan L, Gianaros PJ, Erickson KI. Effects of a laboratory-based aerobic exercise intervention on brain volume and cardiovascular health markers: protocol for a randomised clinical trial. BMJ Open. 2023 Nov 15;13(11):e077905. doi: 10.1136/bmjopen-2023-077905. PMID 37968003

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aerobic Exercise Group | Physical Activity & Health Information Group
Started | 64 | 66
Completed | 41 | 41
Not Completed | 23 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise Group | Physical Activity & Health Information Group | Total
Number analyzed (Participants) | 64 | 66 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.55 (10.48) | 40.98 (9.40) | 41.26 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 45 | 88
  Male | 21 | 21 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 59 | 64 | 123
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 5 | 16
  White | 42 | 49 | 91
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 2 | 1 | 3
VO2peak [Mean (Standard Deviation); unit: mL/kg/min] — Peak oxygen uptake (VO2peak) is the highest VO2 value obtained during the maximal test and represents the measure of cardiorespiratory fitness used in this study.
  mL/kg/min | 26.85 (6.60) | 30.23 (6.93) | 28.57 (6.95)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hippocampal Volume
Description: Magnetic Resonance Imaging (MRI) will be used to measure the structure of the brain. Segmentation algorithms applied to structural MRI images will be used to compute the volume of the hippocampus in particular, which will be evaluated for change over the course of the trial.
Time Frame: Baseline & 12 months
Population: All randomized participants were included in intention-to-treat (ITT) analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm^3
Arm/Group | Aerobic Exercise Group | Physical Activity & Health Information Group
Number analyzed (Participants) | 64 | 66
mm^3 | -15.4 [-79.3 to 48.4] | -49.9 [-112.8 to 13]

2. Secondary Outcome: Change in Systolic Blood Pressure Responses to Behavioral Tasks
Description: Average systolic blood pressure will be computed during a resting baseline period and during the performance of two behavioral tasks, (1) a Stroop color-word interference task and (2) a multi-source interference task. Mean baseline levels of systolic blood pressure will be subtracted from mean levels averaged across the two tasks to compute response scores, and changes in task-response scores will be evaluated over the course of the trial.
Time Frame: Baseline & 12 months
Population: Randomized participants who had baseline systolic blood pressure measures available were included in intention-to-treat (ITT) analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Aerobic Exercise Group | Physical Activity & Health Information Group
Number analyzed (Participants) | 55 | 62
mmHg | -0.932 [-3.7 to 1.836] | -3.519 [-6.2 to -0.835]

3. Secondary Outcome: Change in Heart Rate Variability (HRV)
Description: Heart rate variability will be computed from inter-beat intervals derived from electrocardiographic recordings while participants rest in the seated position. Average heart rate variability values from the recording period will be assessed for their change over the trial. Here, we report the natural log-transformed variance of high-frequency (HF) heart rate variability.
Time Frame: Baseline & 12 months
Population: Randomized participants who had heart rate variability measures available at baseline were included in intention-to-treat (ITT) analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: ln[ms²]
Arm/Group | Aerobic Exercise Group | Physical Activity & Health Information Group
Number analyzed (Participants) | 61 | 62
ln[ms²] | 0.0022 [-0.257 to 0.261] | -0.2035 [-0.472 to 0.065]

4. Other Pre Specified Outcome: Change in fMRI
Description: Changes in task invoked activity will be measured during an emotion regulation task.
Time Frame: Baseline & 12 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Reappraisal and Suppression Scores
Description: Participants will complete the Emotion Regulation Questionnaire (ERQ). They rate how strongly they agree with 10 statements and emotion regulation abilities are calculated by their responses. A minimum score would be 10 and a maximum score would be 70, with 70 indicating superior emotion regulation abilities.
Time Frame: Baseline, 6-month (if applicable) & 12 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Perceived Stress Scale (PSS)
Description: This will be calculated via the PSS 4-item scale. Scores are calculated by averaging responses from 10 questions with a minimum score of 0 and a maximum score of 40. 40 indicates more stress.
Time Frame: Baseline, 6-month (if applicable) & 12 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Self-esteem
Description: Participants will complete a questionnaire related to self-esteem via the Rosenberg Self Esteem Scale. All items are answered using a 4-point Likert scale format ranging from strongly agree to strongly disagree. Sum scores for all 10 items are calculated with items 2, 5, 6, 8, 9 being reverse scored. Higher scores indicate higher self-esteem.
Time Frame: Baseline, 6-month (if applicable) & 12 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Blood Pressure
Description: An average systolic blood pressure (SBP) will be calculated for an average over all baseline, 6-month (if applicable) and 12-month visits.
Time Frame: Baseline, 6-month (if applicable), & 12 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Cardiorespiratory Fitness
Description: Fitness is assessed by maximal graded exercise testing. Oxygen uptake (VO2) will be measured from expired air samples taken at 15s intervals until a peak VO2, the highest VO2, is attained at the point of test termination due to symptom limitation and/or volitional exhaustion.
Time Frame: Baseline, 6-month (if applicable), & 12-month
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Fasting Glucose.
Description: Blood will be drawn at 3 time points throughout the intervention starting at baseline to measure changes in fasting glucose.
Time Frame: Baseline, 6-month (if applicable) & 12 month
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Insulin Resistance.
Description: Blood will be drawn at 3 time points throughout the intervention starting at baseline to measure changes in insulin resistance.
Time Frame: Baseline, 6-month (if applicable) & 12 month
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Mediation
Description: The outcome will be measured by whether the statistical mediation model that contains brain and peripheral physiological mediators is significant. By definition such a model must contain multiple outcome variables, but the outcome here isn't a measurable outcome but rather whether the statistical model with these variables reaches statistical significance.
Time Frame: Baseline, 6 month (if applicable) and 12 month.
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Heart Rate
Description: An average heart rate will be calculated for an average over all baseline, 6-month (if applicable) and 12-month visits.
Time Frame: Baseline, 6-month (if applicable), & 12 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Daily Life Ecological Monitoring Assessment (EMA)
Description: Participants will complete several questions on a smart phone at various times throughout the day based on a prompt to learn more about positive and negative affect. An average positive and negative affect score will be computed.
Time Frame: Baseline & 12 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in Daily Life SBP Reactivity
Description: Participants will have their blood pressure taken while answering questions about daily stressors and an average SBP score will be computed over the course of the wear period.
Time Frame: Baseline & 12 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in Negative and Positive Affect
Description: This will be calculated via scores from the Positive and Negative Affect Scale. Scores can range from 1 to 100, with 1 meaning less positive affect and 100 meaning more positive affect.
Time Frame: Baseline & 12 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in Baroreflex Sensitivity (BRS)
Description: Participants will have electrodes placed on their skin to record an EKG as well as a blood pressure cuff on their arm. BRS will be derived in part from the EKG signal.
Time Frame: Baseline & 12 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change in Pulse Wave Velocity (PWV)
Description: Participants will have electrodes placed on their skin to record an EKG as well as a blood pressure cuff on their arm. PWV will be derived in part from the EKG signal.
Time Frame: Baseline & 12 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change in Vasodilation (Reactive Hyperemia)
Description: Participants will have electrodes placed on their skin to record an EKG as well as a blood pressure cuff on their arm. Vasodilation (reactive hyperemia) will be derived in part from the EKG signal.
Time Frame: Baseline & 12 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Change in Brain Activity
Description: MRI will be used to measure changes in brain activity including task invoked activation patterns.
Time Frame: Baseline & 12 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Change in Resting State Connectivity
Description: MRI will be used to measure changes in functional connectivity during rest.
Time Frame: Baseline & 12 months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Change in Cortical Thickness.
Description: MRI will be used to measure cortical thickness. Measured in mm3.
Time Frame: Baseline & 12 months
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Change in Cortical Volume.
Description: MRI will be used to measure cortical volume. Measured in mm3.
Time Frame: Baseline & 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Aerobic Exercise Group | Physical Activity & Health Information Group
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/64 | 0/66
Other Adverse Events (participants affected / at risk) | 6/64 | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Exercise Group (N=64) | Physical Activity & Health Information Group (N=66)
Tumor (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Exercise Group (N=64) | Physical Activity & Health Information Group (N=66)
Cardiovascular (Vascular disorders) | 1 | 0
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 | 0 — Bone fracture, back pain, ankle sprain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT03841669/Prot_SAP_000.pdf